CLINICAL TRIAL: NCT03730311
Title: Phase Ib, Single-Centre, Placebo-Controlled Randomised Study of Safety, Tolerability and Pharmacokinetics of Elpida in Healthy HIV-Uninfected Volunteers
Brief Title: Phase Ib Study of Safety, Tolerability and Pharmacokinetics of Elpida Once Weekly in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HIV-VM1500-11
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — elsulfavirine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Elpida 120 mg once weekly (Experimental): elsulfavirine 120mg or placebo orally once weekly for 4 weeks
  Interventions: Drug: Elpida; Drug: placebo
- Elpida 200 mg once weekly (Experimental): elsulfavirine 200mg or placebo orally once weekly for 4 weeks
  Interventions: Drug: Elpida; Drug: placebo
- Elpida 280 mg once weekly (Experimental): elsulfavirine 280mg or placebo orally once weekly for 4 weeks
  Interventions: Drug: Elpida; Drug: placebo

INTERVENTIONS:
Drug: Elpida — elsulfavirine, capsules
  Other Names: elsulfavirine; VM-1500; VM1500
Drug: placebo — placebo

SUMMARY:
A randomized, placebo-controlled, once weekly dose for four weeks, double blind study in Healthy HIV-Uninfected Volunteers. Each of 3 consequent groups (120 mg, 200 mg and 280mg) enrolls 6 active and 2 placebo subjects.

DETAILED DESCRIPTION:
The study aims to assess safety, tolerability and PK of once weekly administration of Elpida in different doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females aged between 18-40 years.
2. Willing and able to complete all study procedures, visits and restrictions.
3. Capable of giving written informed consent.
4. Has been determined healthy by medical history, physical and vital signs examinations.
5. Has normal results for the following screening tests: complete blood count (CBC), sodium, potassium, blood urea nitrogen (BUN), serum creatinine, fasting blood sugar (FBS), creatine kinase, total calcium, cholesterol, triglyceride, total protein, total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) and urinalysis.
6. Females of reproductive potential (defined as women who have not been postmenopausal for at least 24 consecutive months [i.e., who have had menses within the preceding 24 months], or women who have not undergone surgical sterilization; specifically hysterectomy, salpingotomy, bilateral oophorectomy, and/or tubal ligation), must have a negative serum or urine pregnancy test with a sensitivity of at least 40 mIU/mL at Screening and prior to drug dosing on Day 1.
7. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). If participating in sexual activity that could lead to pregnancy, the participant must agree to use two reliable methods of contraception simultaneously while receiving study treatment and for 6 months after stopping study drug. Subjects must either be abstinent or a combination of TWO of the following methods MUST be used appropriately:

   * Condoms (male or female) with or without a spermicidal agent;
   * Diaphragm or cervical cap with spermicide;
   * Intrauterine device (IUD);
   * Hormonal-based contraception. Participants who are not of reproductive potential (women who have been postmenopausal for at least 24 consecutive months or have undergone hysterectomy, salpingotomy, bilateral oophorectomy, and/or tubal ligation or men who have documented azoospermia) are eligible without requiring the use of contraceptives. Acceptable documentation of sterilization, menopause or male partner's azoospermia must be provided; serum follicle stimulating hormone (FSH) measurement can be used to document menopausal range.

Exclusion Criteria:

1. Hepatic or kidney disorders or any other disease or disorder which may in the opinion of the Investigator interfere with the results of the study or threaten the health of volunteers.
2. Clinically significant ECG abnormality according to ECG exam at Screening, subject's medical history or family history judged by the Investigator that the presence of, or an increased risk of cardiac abnormality.
3. Positive result for HIV, HCV or HBV at Screening.
4. Positive result for illicit drugs screen (opiates, amphetamines, cannabinoids or cocaine) or alcohol screen at Screening.
5. Active alcohol or and/or drug abuse that, in the opinion of the site investigator, would interfere with adherence to study requirements.
6. Received the excluded medications (as shown in Appendix 3) within 14 days or 28 days prior to the first dose of study drug, or within the 5 half-lives of individual medication, whichever is longer.
7. Participated in a clinical study and received any investigational drug or vaccine or medical device within 90 days prior to the first dose of study drug.
8. Pregnancy or breast feeding, male partners of pregnant females. Inability to understand the Protocol or follow its instructions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | 36 days
  Incidence of AEs and SAEs

SECONDARY OUTCOMES:
elsulfavirine plasma concentration | 36 days
  elsulfavirine plasma concentration
VM1500A plasma concentration | 36 days
  active metabolite plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Somruedee Chatsiricharoenkul, Assoc. Prof., MD, Principal Investigator — Siriraj Hospital Bangkok, Thailand
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided